CLINICAL TRIAL: NCT03800121
Title: Study of Exosomes in Monitoring Patients With Sarcoma (EXOSARC)
Acronym: EXOSARC
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: INSERM UMR1231 Lipids Nutrition Cancer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-A01393-52
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Sarcoma
Keywords: exosomes
MeSH Terms: conditions — Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Localized sarcoma with neoadjuvant chemotherapy: In total, several blood tests specific to the EXOSARC study will be necessary:
  * A first blood test of 7 mL during the initial assessment (inclusion)
  * Then four blood samples of 32mL distributed over 6 months
  Interventions: Biological: Blood samples
- Metastatic or locally advanced sarcoma: In total, several blood tests specific to the EXOSARC study will be necessary :
  * A first blood of 7 mL during the initial assessment (inclusion)
  * Then three blood samples of 32 mL distribuated over 3 months
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Localized sarcoma group : 1 blood sample during inclusion (7 ml) + 1 blood sample before surgery (32 ml) + 1 blood sample 1 month after surgery (32 ml) + 1 blood sample 3 month after surgery (32 ml) + 1 blood sample 6 month after surgery (32 ml)
  Metastatic sarcoma group : 1 blood sample during inclusion (7 ml) + 1 blood sample during chemotherapy cure 1 (32 ml) + 1 blood sample during chemotherapy cure 3 (32 ml) + 1 blood sample during chemotherapy cure 6 (32 ml)
  Other Names: Localized sarcoma; Metastatic sarcoma

SUMMARY:
Sarcomas are rare cancers with a high risk of metastatic progression and a major pejorative factor with respect to patient survival. The estimation of the metastatic risk of sarcomas is very complex given the histological heterogeneity of this entity. It is therefore essential that, at diagnosis, a reliable evaluation of this metastatic potential be made, in order to adapt the therapeutic strategy as well as possible.

It has recently been discovered that sarcomas secrete many exosomes that appear to play an important role in tumorogenesis, growth, tumor progression and the onset of metastases. They contain many proteins and nucleic acids (DNA, RNA, microRNA), reflecting the characteristics of the tumor. It has been shown that the amount of exosomes can be correlated with the grade of malignancy of the tumor. Present in the blood, exosomes offer the possibility of non-invasively analyzing the molecular information of the cancer cell. As a result, the study of serum exosomes derived from sarcomas has a high potential as a liquid biopsy to evaluate cancer pathogenesis, progression, and treatment efficacy.

The purpose of this study is to demonstrate in patients with sarcomas that exosomes can be used to monitor their disease and be used as a predictor of the risk of recurrence.

DETAILED DESCRIPTION:
The main objective of this pilot study is to quantify exosomes and analyze their protein and RNA content in patients with sarcoma with disease:

* localized before and after treatment with surgery,
* localized for which neoadjuvant chemotherapy is being considered
* metastatic or locally advanced cancer before and after treatment with first-line chemotherapywhich may include neoadjuvant therapy

The secondary objectives are:

1. Determine whether the initial exosome concentration and the protein and RNA profile they contain vary with the localized or metastatic stage of the disease.
2. Determine if the exosome concentration as well as the protein and RNA profile they contain varies after treatment.
3. Determine if the initial exosome concentration (at T0) is associated with a response to treatment.
4. Determine whether the change in exosome concentration before and after treatment is associated with a response to treatment.
5. Identify a protein marker or RNA associated with a treatment response (marker present at T0 or occurring during follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women newly diagnosed with localized, metastatic or locally advanced soft tissue sarcoma
2. Previous treatment of the disease with chemotherapy, radiotherapy or surgery is allowed if it has been completed for more than 12 months at the time of inclusion.
3. For metastatic or locally advanced (inoperable) sarcoma, patients for whom first-line metastatic chemotherapy is indicated.
4. Age ≥18 years
5. Affiliation to a social security scheme
6. Patients who signed informed consent to participate in the study

Exclusion Criteria:

Patients who meet at least one of the following criteria will not be eligible:

1. Patient with another synchronous tumor,
2. Patient with sarcoma in irradiated territory
3. Patient with a history of cancer other than sarcoma in the 5 years preceding the diagnosis of sarcoma
4. Patient unable to undergo medical follow-up for geographical, social or psychological reasons,
5. Person benefiting from a protection system for adults (including guardianship and trusteeship),
6. Serology HIV and / or HBV and / or HCV positive.
7. Pregnant or lactating woman.
8. Patients unable to understand, read and / or sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft tissue sarcoma
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
concentration of exosomes in blood | up to 6 months after inclusion
  blood samples

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vautrot V, Hervieu A, Bertaut A, Charon-Barra C, Naiken I, Causseret S, Chaigneau L, Desmoulins I, Rederstoff E, Isambert N, Gobbo J. Small Extracellular Vesicles as Biomarkers in Sarcoma Follow-Up: Protocol for a Prospective, Multicentric Pilot Study. JMIR Res Protoc. 2025 Sep 9;14:e63718. doi: 10.2196/63718. PMID 40925003